CLINICAL TRIAL: NCT00787891
Title: A Multi-Center, Double-Blind, Parallel-Group Study to Evaluate Short-term Safety and Efficacy and Long-Term Maintenance of Two Dose Levels of Rabeprazole Sodium Delayed-Release Pediatric Bead Formulation in 1- to 11-Year Old Pediatric Subjects With Endoscopically Proven GERD
Brief Title: A Study of the Safety and Effectiveness of Rabeprazole for the Treatment of Gastroesophageal Reflux Disease (GERD) in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014833; RABGRD3003 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease (GERD); Erosive Gastroesophageal Reflux Disease; Ulcerative Gastroesophageal Reflux Disease; Endoscopy; Pediatrics; Rabeprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rabeprazole 0.5 mg/kg (Experimental): rabeprazole 0.5mg/kg once daily for 12 weeks plus option for F/u another 24 weeks
  Interventions: Drug: rabeprazole
- Rabeprazole 1.0 mg/kg (Experimental): rabeprazole 1.0 mg/kg once daily for 12 weeks plus option for F/u another 24 weeks
  Interventions: Drug: rabeprazole

INTERVENTIONS:
Drug: rabeprazole — 0.5mg/kg once daily for 12 weeks plus option for F/u another 24 weeks
  Arms: Rabeprazole 0.5 mg/kg
Drug: rabeprazole — 1.0 mg/kg once daily for 12 weeks plus option for F/u another 24 weeks
  Arms: Rabeprazole 1.0 mg/kg

SUMMARY:
The purpose of the study is to access the effectiveness and safety of oral rabeprazole in the treatment of acid-related disorders in pediatric patients, focusing specifically on the manifestation of GERD (symptomatic and erosive types).

DETAILED DESCRIPTION:
This is a randomized, double-blind study that consists of two parts. In Part 1, the study will consist of 3 phases: a 14-day screening phase, a double-blind treatment phase of 12 weeks comparing two doses of study drug (0.5 mg/kg or 1.0 mg/kg groups based on patient's body weight), and an end-of-study or early withdrawal phase followed by Part 2, which consists a of double-blind treatment continuation for patients who have achieved healing during the short-term double-blind treatment phase. The double-blind maintenance treatment phase lasts for not more than 24 weeks and is concluded by an end-of-study/early withdrawal visit. During Part 1, patients will be screened and the diagnosis of erosive and non-erosive Gastroesophageal Reflux Disease (GERD) will be made based on clinical symptoms and confirmed by endoscopy/histology after a biopsy. Patients enrolled in the study will receive study drug once daily for 12 weeks. Each day, the parent/caregiver will record the presence and severity of pre-specified GERD symptoms. At Weeks 4 and 8, the investigator will evaluate the response to treatment by assessment of the GERD symptoms. At Week 12, the investigator will perform an endoscopy of the esophagus with a biopsy to confirm that histological healing has occurred. If a patient continues, additional study drug will be dispensed (at the same dose taken during the short-term double-blind treatment phase) and the patient will be scheduled to return every 8 weeks until study drug is discontinued at Week 24 (Part 2) of the double-blind maintenance treatment phase. At the final visit of the maintenance treatment phase Week 24 (Part 2), assessments including an endoscopy of the esophagus with a biopsy be performed for each patient. Assessments of effectiveness include endoscopic and histological grading of biopsy samples, GERD symptom and severity score (symptoms and severity rated daily by the parent/caregiver in an electronic diary), overall GERD symptom relief, Clinical Global Impression of Improvement (CGI-I) score, and the Global Treatment Satisfaction Score. Safety assessments will include the monitoring of concomitant therapies and adverse events throughout the study, clinical laboratory testing (including hematology, clinical chemistry, urinalysis), vital signs, and physical examination including height, weight, and Tanner staging. Oral rabeprazole 2.5 capsules or 5 mg capsules, given once daily at a dose of 0.5 mg/kg or 1.0 mg/kg; short-term treatment phase is 12 weeks; long-term maintenance treatment phase is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of at least 1 Gastroesophageal Reflux Disease (GERD) symptom within 3 months of screening
* Positive esophagogastroduodenoscopy
* Signed informed consent
* Female patients (if menstruating) must be practicing birth control

Exclusion Criteria:

* Patients with history of esophagitis
* Patients who have milk protein allergy
* Patients who have taken Proton Pump Inhibitors or H2-blockers within 3 days
* Patients who have taken sucralate or any medication that affects gastrointestinal motility
* Patients with H. pylori
* Patients with lab values outside the normal age appropriate range
* Patients who have participated in another trial within 30 days before screening
* Patients with allergies to Proton Pump Inhibitors

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Haddad I, Kierkus J, Tron E, Ulmer A, Hu P, Sloan S, Silber S, Leitz G. Efficacy and safety of rabeprazole in children (1-11 years) with gastroesophageal reflux disease. J Pediatr Gastroenterol Nutr. 2013 Dec;57(6):798-807. doi: 10.1097/MPG.0b013e3182a4e718. PMID 23863328

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, 108 patients completed the 12-week phase (Part 1) and were counted for the primary outcome measure (OM). Patients with healing at Week 12 had the option to continue the treatment for 24 weeks. Among the 87 with healing, 64 enrolled into Part 2. Only 52 had the primary efficacy endpoint available and were included in the primary OM.
Groups:
- Rabeprazole 0.5 mg/kg; Rabeprazole 1.0 mg/kg: Pediatric micro-bead formulation of rabeprazole sodium orally administered.
Period: Short-term Double-blind Phase (Part 1)
Arm/Group | Rabeprazole 0.5 mg/kg | Rabeprazole 1.0 mg/kg
Started | 65 | 62
Completed | 55 | 53
Not Completed | 10 | 9
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Other | 0 | 2
Period: Maintenance Double-blind Phase (Part 2)
Arm/Group | Rabeprazole 0.5 mg/kg | Rabeprazole 1.0 mg/kg
Started | 33 | 31
Completed | 26 | 24
Not Completed | 7 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Non-Compliance With Study Drug | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabeprazole 0.5 mg/kg | Rabeprazole 1.0 mg/kg | Total
Number analyzed (Participants) | 65 | 62 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 65 | 62 | 127
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 5.9 (3.49) | 5.4 (3.26) | 5.7 (3.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 56
  Male | 34 | 37 | 71
Baseline BMI [Mean (Standard Deviation); unit: kg/cm2] | 17.5 (4.08) | 16.8 (3.11) | 17.2 (3.64)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Healing by Week 12 (Short-term Double-blind Treatment Phase)
Description: Healing is defined as macroscopically normal esophageal mucosa or histologic normal esophageal mucosa.
Time Frame: 12 weeks
Population: Intention to Treat (ITT) analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Rabeprazole Sodium 0.5 mg/kg; Rabeprazole Sodium 1.0 mg/kg: Pediatric micro-bead formulation of rabeprazole sodium orally administered.
Arm/Group | Rabeprazole Sodium 0.5 mg/kg | Rabeprazole Sodium 1.0 mg/kg
Number analyzed (Participants) | 55 | 53
Percentage of participants | 78 [67 to 89] | 83 [73 to 93]

2. Primary Outcome: The Percentage of Patients With Healing by Week 36 (Double-blind Maintenance Treatment Phase)
Description: Healing is defined as macroscopically normal esophageal mucosa or histologic normal esophageal mucosa.
Time Frame: 36 weeks
Population: Intention to Treat (ITT) analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Rabeprazole Sodium 0.5 mg/kg | Rabeprazole Sodium 1.0 mg/kg
Number analyzed (Participants) | 26 | 26
Percentage of patients | 92 [82 to 100] | 88 [76 to 100]

3. Secondary Outcome: The Change From Baseline in the Hetzel and Dent Endoscopic Classification Grade Score (Short-term Double-blind Treatment Phase)
Description: The Hetzel and Dent Classification grades range from 0 (normal esophageal mucosa, no abnormalities noted) to 4 (deep ulcers anywhere in the esophagus or ulceration of more than half of the esophageal mucosa). Higher observed scores indicate more serious condition. For change of baseline, a score of 0 indicates no change; a positive score indicates the condition is worsening, while a negative score indicates an improvement.
Time Frame: Baseline, Week 12
Population: Intention to Treat (ITT) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rabeprazole Sodium 0.5 mg/kg | Rabeprazole Sodium 1.0 mg/kg
Number analyzed (Participants) | 55 | 53
Scores on a scale | -1.3 (0.85) | -1.0 (0.81)

4. Secondary Outcome: The Change From Baseline in the Total GERD Symptom and Severity Score (Short-term Double-blind Treatment Phase)
Description: The gastroesophageal reflux disease (GERD) symptom and severity scale measures the frequency (0= Never; 1= 1-2 times; 2= 3-4 times; 3= 5-6 times; 4= 7 or more times) and the severity (1= Mild; 2= Moderate; 3=Severe) of GERD symptoms. The score is defined as the sum of the frequency (0-4) and severity (1-3) of that symptom. The total score is the sum of the scores of all the symptoms and ranges from 12 to 84. Higher scores indicate more serious condition. For change from baseline, 0 indicates no change; a positive score indicates worsening, while a negative score indicates improvement.
Time Frame: Baseline, Week 12
Population: Intention to Treat (ITT) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rabeprazole Sodium 0.5 mg/kg | Rabeprazole Sodium 1.0 mg/kg
Number analyzed (Participants) | 61 | 59
Scores on a scale | -11.5 (11.70) | -8.5 (9.75)

5. Secondary Outcome: The Change From Baseline in the Hetzel and Dent Endoscopic Classification Grade Score (Double-blind Maintenance Treatment Phase)
Description: as for outcome 3
Time Frame: Baseline, Week 36
Population: Intention to Treat (ITT) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rabeprazole Sodium 0.5 mg/kg | Rabeprazole Sodium 1.0 mg/kg
Number analyzed (Participants) | 26 | 26
Scores on a scale | 0.2 (0.49) | 0.2 (0.54)

6. Secondary Outcome: The Change From Baseline in the Total GERD Symptom and Severity Score (Double-blind Maintenance Treatment Phase)
Description: as for outcome 4
Time Frame: Baseline, Week 36
Population: Intention to Treat (ITT) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rabeprazole Sodium 0.5 mg/kg | Rabeprazole Sodium 1.0 mg/kg
Number analyzed (Participants) | 32 | 29
Scores on a scale | -2.9 (4.82) | -1.4 (9.59)

ADVERSE EVENTS:
Groups:
- Rabeprazole 0.5 mg/kg (Short-term Double-blinde Phase); Rabeprazole 1.0 mg/kg (Short-term Double-blinde Phase); Rabeprazole 0.5 mg/kg (Double-blind Maintenance Phase); Rabeprazole 1.0 mg/kg (Double-blind Maintenance Phase: Pediatric micro-bead formulation of rabeprazole sodium orally administered.
Arm/Group | Rabeprazole 0.5 mg/kg (Short-term Double-blinde Phase) | Rabeprazole 1.0 mg/kg (Short-term Double-blinde Phase) | Rabeprazole 0.5 mg/kg (Double-blind Maintenance Phase) | Rabeprazole 1.0 mg/kg (Double-blind Maintenance Phase
Serious Adverse Events (participants affected / at risk) | 5/65 | 1/62 | 2/33 | 3/31
Other Adverse Events (participants affected / at risk) | 47/65 | 47/62 | 18/33 | 21/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole 0.5 mg/kg (Short-term Double-blinde Phase) (N=65) | Rabeprazole 1.0 mg/kg (Short-term Double-blinde Phase) (N=62) | Rabeprazole 0.5 mg/kg (Double-blind Maintenance Phase) (N=33) | Rabeprazole 1.0 mg/kg (Double-blind Maintenance Phase (N=31)
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Partial Seizures with Secondary Generalisation (Nervous system disorders) | 0 | 0 | 1 | 0
Conversion Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole 0.5 mg/kg (Short-term Double-blinde Phase) (N=65) | Rabeprazole 1.0 mg/kg (Short-term Double-blinde Phase) (N=62) | Rabeprazole 0.5 mg/kg (Double-blind Maintenance Phase) (N=33) | Rabeprazole 1.0 mg/kg (Double-blind Maintenance Phase (N=31)
Abdominal Pain (Gastrointestinal disorders) | 7 | 8 | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 8 | 10 | 4 | 3
Pyrexia (General disorders) | 8 | 5 | 0 | 3
Bronchitis (Infections and infestations) | 1 | 2 | 1 | 0
Croup Infectious (Infections and infestations) | 1 | 0 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Localised Infection (Infections and infestations) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 2 | 1
Otitis Media (Infections and infestations) | 3 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 3 | 1 | 1 | 1
Pharyngitis Streptococcal (Infections and infestations) | 1 | 1 | 2 | 1
Rhinitis (Infections and infestations) | 3 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 2 | 3 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 4 | 4 | 4
Viral Infection (Infections and infestations) | 1 | 2 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 4 | 7 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 3 | 0 | 0
Eustachian Tube Obstruction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 2 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Eosinophilic Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Acute Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis Infective (Infections and infestations) | 0 | 1 | 0 | 0
Coxsackie Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 1 | 0
Molluscum Contagiosum (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Asthma Exercise Induced (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Menarche (Social circumstances) | 0 | 1 | 0 | 0
Suture Insertion (Surgical and medical procedures) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Atopy (Immune system disorders) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Beta 2 Microglobulin Urine Increased (Investigations) | 0 | 0 | 1 | 0
Blood Iron Decreased (Investigations) | 0 | 0 | 0 | 1
Serum Ferritin Decreased (Investigations) | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Febrile Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Breast Mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Fungal Oesophagitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis Rotavirus (Infections and infestations) | 0 | 0 | 0 | 1
Rash Pustular (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less